CLINICAL TRIAL: NCT06228547
Title: Women's Experience of Premature Ovarian Insufficiency (POI) Diagnosis: Update on Actual Practices and Patient's Follow up
Acronym: EMPOIHER
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/24
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Premature Ovarian Insufficiency
Keywords: Premature ovarian insufficiency; diagnosis; patient satisfaction; gynecological follow-up; hormone replacement therapy
MeSH Terms: conditions — Primary Ovarian Insufficiency; Disease; Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- POI: Woman aged 18 years and older, diagnosed with POI following ESHRE 2016 criteria
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Standardized questionnaire specifically made for the study. The interview lasts approximately 15 minutes. The form gathers baseline characteristics of the patients such as socio-demographic information, symptoms, lifestyle factors and gynecological history. The questionnaire focuses also on the manner in which the diagnosis was revealed to the patient and their experience of this disclosure. Lastly, the questionnaire includes items issued from French practice guidelines concerning etiological investigations, fertility assessment, osteoporotic and cardiovascular complications, HRT use, and residual symptoms

SUMMARY:
Premature ovarian insufficiency (POI) affects 2,8 to 3,5% of women before the age of 40. Previous foreign studies revealed that only half of POI disclosures occurred during a medical consultation and that the diagnosis was often discussed in less than 5 minutes. As a result, most of patients felt a lack of information, and consequently sought data on the internet. None of these studies were conducted in France. The aim of this study is to analyze current practices related to POI diagnosis and to assess women's satisfaction

DETAILED DESCRIPTION:
POI is defined by the association of 1 clinical and 1 biological criterion: amenorrhea or spaniomenorrhea of > 4 months with onset before 40 year of age, and elevated follicle-stimulating hormone (FSH) > 25 IU/L on 2 assays at > 4 weeks' interval, associated with low estradiol level. This condition affects approximately 2% of young women.

POI can first lead to infertility and various symptoms caused by a lack of estrogens. Thus, patients may experience vaso-motor flushes, genitourinary syndrome, sleep disturbance, humor disorder, decrease libido and dyspareunia. After several years, POI can lead to osteoporosis, increased cardiovascular risk, and dementia. The administration of hormone replacement therapy (HRT) can help prevent these complications. Otherwise, POI may result in psychological repercussions such as anxiety, anger, loss of self-esteem, even depression.

Few studies analyzed POI diagnosis and the way it was perceived by patients. Alzubaidi et al. and subsequently Groff et al. reported that only half of POI notifications occurred during a medical consultation. Moreover, 35% of the consultations lasted less than 5 minutes. Thereby, Singer et al. founds that 68% of women felt inadequately informed. The majority of patients sought additional information on the internet.

No recent study focused on the disclosure of POI diagnosis, and none of the existing studies were conducted in France. The purpose of this study is to analyze the circumstances surrounding POI diagnosis and to evaluate women's experience.

In other ways, in 2016, Bachelot et al. emphasized that after more than 5 years after POI diagnosis, only 61,7% of women were undergoing HRT whereas only 6% had no regular follow-up. Moreover, among the treated patients, 42,6% had already stopped HRT for more than 1 year without any medical recommendation. Therefore, this study aims to examine the association between women satisfaction regarding POI disclosure and their compliance to HRT and medical follow-up

ELIGIBILITY:
Inclusion Criteria:

* woman aged 18 years and older,
* diagnosed with POI following ESHRE 2016 criteria,
* speaking and reading French language,
* woman's oral consent,
* affiliated or beneficiary of health insurance.

Exclusion Criteria:

* iatrogenic POI (surgery, radiotherapy, chemotherapy linked),
* chromosomic POI (Turner Syndrome),
* inability for the woman to understand the nature or risks or significance and implications of the study,
* woman under legal protection

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Woman aged 18 years and older, diagnosed with POI following ESHRE 2016 criteria
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
women's satisfaction | Baseline
  Women's satisfaction regarding POI disclosure will be evaluated using a standardized questionnaire specifically made for this study. Findings will be presented as a score based on 5 questions assessing patient's experience of POI diagnosis (Healthcare provider adjustments to patient's emotional state, speech clarity, information provided, opportunity to ask questions, relevance of the topics discussed based on the patient's concerns). For each question a score from 1 to 4 will be assigned (Very unsatisfied = 1 ; Unsatisfied = 2 ; Satisfied = 3 ; Very satisfied = 4), resulting in a total score ranging from 5 to 20. Patients scoring from 5 to 8 will be categorized as overall very unsatisfied, 9 to 12 as unsatisfied, 13 to 16 as satisfied, and 17 to 20 as very satisfied

SECONDARY OUTCOMES:
Patient's expectations | Baseline
  Patient's expectations regarding POI disclosure
gynecological follow-up | Baseline
  Rate of patients having regular gynecological follow-up
hormone replacement therapy | Baseline
  Percentage of patients undergoing hormone replacement therapy (HRT)
interrupted HRT | Baseline
  Percentage of patients who interrupted HRT for more than one year
bone mineral density evaluation | Baseline
  Percentage of patients who ever had a bone mineral density evaluation
osteoporosis | Baseline
  Prevalence of osteoporosis
cardiovascular risk factor | Baseline
  Prevalence of patients with cardiovascular risk factor(s).
side effects when taking HRT | Baseline
  Prevalence of patients experiencing side effects when taking HRT
residual symptoms of POI | Baseline
  Prevalence of patients with residual symptoms of POI despite HRT
cervical cancer | Baseline
  Percentage of patients who had cervical cancer screening following current guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No